CLINICAL TRIAL: NCT01244334
Title: A Randomized, Masked Multi-center Safety & Efficacy Study of the Effects of Preoperative & Postoperative Cataract Surgery Use of Difluprednate Ophthalmic Emulsion, 0.05% Compared to Prednisolone Acetate Ophthalmic Suspension 1% on Visual Acuity & Corneal Edema.
Brief Title: Study of Difluprednate vs. Prednisolone Acetate on Visual Acuity, and Corneal Edema Following Cataract Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edward J. Holland (Other)
Collaborators: Sirion Therapeutics, Inc. (Industry); Alcon Research (Industry); Parsons Medical Communications (Unknown)
Responsible Party: Sponsor-Investigator, Edward J. Holland, Sponsor Investigator, Cincinnati Eye Institute Northern Kentucky
Organization: Cincinnati Eye Institute Northern Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEMC 5/2009-011
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Cataracts; Corneal Edema; Retinal Structural Change, Deposit and Degeneration; Visual Acuity Reduced Transiently
Keywords: cataract surgery, vision, corneal edema, retinal thickness
MeSH Terms: conditions — Cataract; Corneal Edema | interventions — difluprednate; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Difluprednate Ophthalmic Emulsion 0.05% (Active Comparator)
  Interventions: Drug: Difluprednate ophthalmic emulsion 0.05%
- Prednisolone acetate suspension 0.1% (Active Comparator)
  Interventions: Drug: Prednisolone acetate 1%

INTERVENTIONS:
Drug: Difluprednate ophthalmic emulsion 0.05% — Difluprednate ophthalmic emulsion 0.05%: 29 days total, total of 7 drops prior to surgery, and 3 more following surgery while at the surgery center, then Q2H on day of surgery, then QID for 1 week, then BID for 1 week, then stop.
  Other Names: Durezol
  Arms: Difluprednate Ophthalmic Emulsion 0.05%
Drug: Prednisolone acetate 1% — Prednisolone acetate 1% : 29 days total, total of 7 drops prior to surgery, and 3 more following surgery while at the surgery center, then Q2H on day of surgery, then QID for 1 week, then BID for 1 week, then stop.
  Other Names: Prednisolone acetate
  Arms: Prednisolone acetate suspension 0.1%

SUMMARY:
The purpose of this clinical research study is to investigate the efficacy of predosing patients undergoing cataract surgery with the potent corticosteroid difluprednate ophthalmic emulsion 0.05% compared to prednisolone acetate 1% on corneal edema (swelling), and retinal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 21 years of age or older
* Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6-25 days between surgeries.
* Willing and able to administer eye drops and record the times the drops were instilled
* Understand and are willing to sign the Informed Consent form
* Willing to complete the entire course of the study.

Exclusion Criteria:

* Use of an eye medication or drops within 48 hours of the scheduled cataract surgery, other than the study medication or procedural solution required for surgery.
* Known sensitivity to any of the ingredients in the study medications or similar medications.
* Scheduled for 2nd eye cataract surgery earlier than 6 days or longer than 25 days apart.
* Corneal edema in either eye.
* Need for regional or general anesthesia during surgery.
* Complicated cataract surgery, including use of iris hooks or iris stretchers.
* Sight better than 20/100 in only one eye.
* A history of previous intraocular surgery in either eye.
* A history of uveitis, iritis, or intraocular inflammation.
* Macular pathology of the retina.
* Presence of glaucoma.
* Any confirmed or suspected active viral, bacterial, or fungal keratoconjunctival disease.
* History of steroid-related intraocular pressure (IOP) rise in the study eye.
* Lack of an intact corneal epithelium.
* Pupils that do not dilate to more than 5 mm prior to surgery or you require mechanical stretching of your pupil.
* Diabetes mellitus.
* Required use of a systemic steroidal or non-steroidal anti-inflammatory during the study period.
* Doctor has determined the presence of a condition (i.e., UNCONTROLLED systemic disease) or a situation that may put the subject at significant risk, confound the study results or may interfere significantly with your participation in the study.
* Females, who are pregnant, nursing an infant or planning a pregnancy.
* Currently involved in another investigational study or have participated in one within the 30 days prior to entering this study.
* Unable or unwilling to give signed informed consent prior to participation in any study-related procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assess change from Baseline on visual acuity, corneal edema, and retinal thickness at Day 1 | Change from Baseline in visual acuity, corneal edema, and retinal thickness at Day 1

SECONDARY OUTCOMES:
Assess change from Baseline on visual acuity, corneal edema, and retinal thickness at Day 15 | change from Baseline on visual acuity, corneal edema, and retinal thickness at Day 15

OTHER OUTCOMES:
change from Baseline on visual acuity, corneal edema, and retinal thickness at Day 30 | change from Baseline on visual acuity, corneal edema, and retinal thickness at Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Holland, MD, Principal Investigator — Cincinnati Eye Institute; Eric D Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island; Kerry S Solomon, MD, Principal Investigator — Carolina Eyecare
Locations (3):
- United States (3):
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Carolina Eyecare, Mt. Pleasant, South Carolina

REFERENCES:
- [Derived] Donnenfeld ED, Holland EJ, Solomon KD, Fiore J, Gobbo A, Prince J, Sandoval HP, Shull ER, Perry HD. A multicenter randomized controlled fellow eye trial of pulse-dosed difluprednate 0.05% versus prednisolone acetate 1% in cataract surgery. Am J Ophthalmol. 2011 Oct;152(4):609-617.e1. doi: 10.1016/j.ajo.2011.03.018. Epub 2011 Jun 25. PMID 21704965